CLINICAL TRIAL: NCT03897647
Title: Use of POC Pocket Ultrasound in the Estimation of Left and Right Atrial Pressures
Acronym: POCUSP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively closed by the IRB
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-8253
Record Dates: First submitted 2018-05-24; First posted 2019-04-01 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Heart Failure; Acute Decompensated Heart Failure
Keywords: echocardiography; pulmonary artery catheter; point of care ultrasound
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- POCUS Patients (Experimental): A bedside echocardiogram will be taken using a point-of-care pocket ultrasound (General Electric (GE) Vscan). Central venous pressure (right atrial pressure) and pulmonary capillary wedge pressure (left atrial pressure) will be collected from pulmonary artery catheters.
  Interventions: Device: General Electric (GE) VScan

INTERVENTIONS:
Device: General Electric (GE) VScan — This is a small, point-of-care, hand-held device used for ultrasound (POCUS). It uses sound waves to generate images without using any radiation.

SUMMARY:
This study will assess the reliability of POC ultrasound in estimating right and left atrium pressures in patients with acute decompensated heart failure. This study will compare hemodynamic measurements obtained from pulmonary artery catheters with those estimated from POC ultrasound using inferior vena cava (IVC) measurements and the presence of atrial septal bulge.

DETAILED DESCRIPTION:
For those patients admitted to the CCU who have pulmonary artery catheters placed by the primary team as part of their medical care, the investigators will collect hemodynamic data from their pulmonary artery catheters and echocardiographic data. Echocardiographic and hemodynamic data obtained from pulmonary artery catheters will be simultaneously collected at baseline (within 24 hours of catheter placement) and after 24 and 48 hours of intensive medical therapy if the pulmonary artery catheter is still in place at those times. The placement of the pulmonary artery catheter and the taking of hemodynamic measurements from the catheter will be done as per the primary medical team. The research team will not place any pulmonary artery catheters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced systolic heart failure (as defined by left ventricular ejection fraction of less than or equal to 35% and New York Heart Association Class III to IV symptoms) who are admitted to the CCU and require hemodynamic monitoring with a Swan-Ganz catheter.

Exclusion Criteria:

* Patients supported by mechanical ventilation (intubation or positive pressure ventilation)
* Patients requiring temporary mechanical circulatory support devices (intra-aortic balloon pump, Impella, CentriMag, extracorporeal membrane oxygenation)
* Patients requiring permanent mechanical circulatory support devices (right or left ventricular assist devices)
* Post-cardiac transplantation patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-31 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Right atrial pressure at baseline | Pressures will be estimated at baseline (within 24 hours of placement of pulmonary artery catheter upon admission to CCU)
  Right atrial pressure is the pressure in one of the chambers of the heart (the right atrium). It reflects the amount of blood returning to the heart. Normal right atrial pressure is 5 to 10 mm Hg. Low pressures indicate that less blood is returning to the heart than normal, higher pressures indicate that more blood is returning to the heart than normal. Higher pressures can occur for example, in patients with heart failure who are fluid overloaded.
Right atrial pressure at 24 hours | Pressures will be estimated 24 hours after baseline
  Right atrial pressure is the pressure in one of the chambers of the heart (the right atrium). It reflects the amount of blood returning to the heart. Normal right atrial pressure is 5 to 10 mm Hg. Low pressures indicate that less blood is returning to the heart than normal, higher pressures indicate that more blood is returning to the heart than normal. Higher pressures can occur for example, in patients with heart failure who are fluid overloaded.
Right atrial pressure at 48 hours | Pressures will be estimated 48 hours after baseline
  Right atrial pressure is the pressure in one of the chambers of the heart (the right atrium). It reflects the amount of blood returning to the heart. Normal right atrial pressure is 5 to 10 mm Hg. Low pressures indicate that less blood is returning to the heart than normal, higher pressures indicate that more blood is returning to the heart than normal. Higher pressures can occur for example, in patients with heart failure who are fluid overloaded.
Left atrial pressure at baseline | Pressures will be estimated at baseline (within 24 hours of placement of pulmonary artery catheter upon admission to CCU)
  Left atrial pressure is the pressure in one of the chambers of the heart (the left atrium). It represents the filling pressure of the left side of the heart before blood is pumped to the rest of the body. Normal left atrial pressure is 6 to 12 mm Hg. In patients with heart failure, the left atrial pressure may be high due to the heart failing to effectively pump blood to the rest of the body.
Left atrial pressure at 24 hours | Pressures will be estimated 24 hours after baseline
  Left atrial pressure is the pressure in one of the chambers of the heart (the left atrium). It represents the filling pressure of the left side of the heart before blood is pumped to the rest of the body. Normal left atrial pressure is 6 to 12 mm Hg. In patients with heart failure, the left atrial pressure may be high due to the heart failing to effectively pump blood to the rest of the body.
Left atrial pressure at 48 hours | Pressures will be estimated 48 hours after baseline
  Left atrial pressure is the pressure in one of the chambers of the heart (the left atrium). It represents the filling pressure of the left side of the heart before blood is pumped to the rest of the body. Normal left atrial pressure is 6 to 12 mm Hg. In patients with heart failure, the left atrial pressure may be high due to the heart failing to effectively pump blood to the rest of the body.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Garcia, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No